CLINICAL TRIAL: NCT03308175
Title: Evaluation of the Effects of Flat and Modified Inclined Fixed Anterior Bite Planes on Mandibular Position in Growing Females With Skeletal Class 2 Malocclusion Due to Mandibular Deficiency and Deep Bite: A Randomized Controlled Trial
Brief Title: Evaluation of the Effects of Flat and Modified Inclined Fixed Anterior Bite Planes on Mandibular Position in Growing Females With Skeletal Class 2 Malocclusion Due to Mandibular Deficiency and Deep Bite
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yomna Elfiky, Resident, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-2017-10-04
Record Dates: First submitted 2017-10-07; First posted 2017-10-12 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2017-10

CONDITIONS: Skeletal Class 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- flat fixed anterior bite plane (Experimental): Bands selection will be done for upper 6s. Alginate impressions taken and molar bands are fitted in place into the impressions. Impressions for upper and lower arches are poured with stone plaster. Mounting on simple hinge articulator will be done.
  Lingual arches (diameter 1 mm) with anterior acrylic bite plates with thickness enough to separate posterior teeth 4mm .
  The acrylic bite planes were in occlusion with the lower anterior teeth and extended sagittally 2-3mm beyond edges of lower incisors.
  Finishing ,polishing and cementation into patient's mouth with glass ionomer cement.
  Interventions: Device: flat fixed anterior bite plane
- modified inclined fixed anterior bite plane (Experimental): In modified inclined fixed anterior bite plane,the modification is that some indentations will be done in the acrylic part where the lower anteriors will fit such that mandible will be held in a more forward position. These indentations will be relieved lingually to overcome it's flaring effect on mandibular incisors .The inclined plane will be 60 degrees to occlusal plane.
  Functional bite will be taken to position the mandible in the proper position forward.
  Bite taken edge-to-edge for appliance construction. Mounting upper and lower casts on simple hinge articulator for construction of modified flat fixed anterior bite plane
  Interventions: Device: modified inclined fixed anterior bite plane

INTERVENTIONS:
Device: flat fixed anterior bite plane — It causes unlocking mandible from deep bite in growing females
  Arms: flat fixed anterior bite plane
Device: modified inclined fixed anterior bite plane — It causes unlocking mandible from deep bite in growing females plus putting the mandible in a more forward position
  Arms: modified inclined fixed anterior bite plane

SUMMARY:
This study will be conducted to see if unlocking mandible from deep bite in growing females by flat fixed anterior bite plane will change mandibular position in skeletal mandibular deficiency and if there is a difference in the change of mandibular position if we assisted the mandible by holding it in a more forward position by modified inclined fixed anterior bite plane .These results will be compared to normal mandibular growth from previous records of a matched control group in the discussion afterthat.

DETAILED DESCRIPTION:
Two groups of patients the first for flat fixed anterior bite plane, the second for modified inclined fixed anterior bite plane.Full records are taken to patients. Then bands selection for upper first molars,impressions for upper arch with bands fitted and impression to lower arch, fabrication of either flat/ modified inclined fixed anterior bite planes and cementation in patient's mouth,evaluation of results after 8 months.

ELIGIBILITY:
Inclusion Criteria:

* (1)Growing females aged 10-13 (2)Skeletal maturational stage: stages 3,4 of the cervical maturational index CVMI.

  (3) low-angle/moderate normal growth pattern (4) Overjet of 4-7 mm as measured from labial surface of upper incisors to labial surface of lower incisors (5)Skeletal class 2 due to mandibular deficiency 77 degrees <SNB> 73 degrees (6) Normal or slightly protruded maxillary base (7) All cases had dental deep bite; with the upper incisors covering more than 50% of the height of the lower incisors.

  (8)Only deep bite cases that required extrusion of posterior teeth.

Exclusion Criteria:1- No syndromic or medically compromised patients 2- No growth disorders 3- No use of other appliances before or during the period of functional treatment

-

Ages: 10 Years to 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2017-11-30 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Change in mandibular position | 8 months
  assessed onCBCT

SECONDARY OUTCOMES:
Maxillary anteroposterior and vertical growth change. | 8 months
  assessed onCBCT
Anteroposterior and vertical dental changes. | 8 months
  assessed onCBCT

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry,Cairo University, Cairo, Egypt